CLINICAL TRIAL: NCT06776315
Title: Examining the Effect of Exercise Training on LncRNA MALAT1 Expression in Asthma Patients
Brief Title: The Effect of Exercise Training on lncRNA Expression in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Fulya Senem Karaahmetoglu, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Asthma_Rehab_lncRNA; 2024/034 (Other Grant/Funding Number: University of Health Sciences Scientific Research Projects Unit)
Record Dates: First submitted 2024-12-13; First posted 2025-01-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Rehabilitation; Pulmonary Rehabilitation; Long Noncoding RNA; Exercise; Asthma
Keywords: Asthma; Pulmonary Rehabilitation; Exercise; Rehabilitation; long noncoding RNA
MeSH Terms: conditions — Motor Activity; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulmonary Rehabilitation Group (PGr) (Active Comparator): In the PGr program, exercises are planned to be performed under the supervision of a remote physiotherapist, 2 days a week with the telerehabilitation method and 1 day as a home-based program by the patient. The exercise program includes aerobic, resistance exercises and respiratory exercises, and patients are followed for 3 months.
  Interventions: Procedure: Standard pulmonary rehabilitation programme
- Pulmonary Rehabilitation Group with Inspiratory Muscle Training (IKE+PGr) (Experimental): In the PGr program, exercises are planned under the supervision of a remote physiotherapist, with the telerehabilitation method 2 days a week and with a program to be done by the patient at home 1 day a week. The exercise program includes aerobics, resistance exercises, respiratory exercises and respiratory muscle strengthening training with a resistive thereshold inspiratory muscle strengthening device, and patients are followed for 3 months.
  Interventions: Device: Resistive threshold inspiratory muscle training device
- Control Group (KGr) (Other): The KGr group will consist of women and men aged between 18-65, who have signed the informed consent form regarding the study, have a BMI <30, are non-smokers, have no known systemic disease, and have FEV1>80, and are age and gender matched to the exercise groups.
  Interventions: Genetic: No intervention

INTERVENTIONS:
Device: Resistive threshold inspiratory muscle training device — In the other arm of the study, respiratory muscle training is performed in addition to the "standard pulmonary rehabilitation program." Respiratory muscle strengthening training is performed with a resistive thereshold inspiratory muscle strengthening device. The exercise is performed at an intensity of 30% of the maximum inspiratory pressure determined by mouth pressure measurement. The exercise is performed in 7 sets, with 2 minutes of work and 1 minute break for a total of 21 minutes.
  Arms: Pulmonary Rehabilitation Group with Inspiratory Muscle Training (IKE+PGr)
Procedure: Standard pulmonary rehabilitation programme — Patients are asked to perform thoracic, diaphragmatic breathing, and lower basal breathing exercises with 10 repetitions. Then, strengthening exercises are performed on the major muscle groups of the upper and lower extremities. In accordance with the resistance training program in the ATS/ERS guidelines for pulmonary rehabilitation, two to four sets of 6-12 repetitions are performed with intensities ranging from 50% to 85% of one maximum repetition, two to three times a week. During the exercises, the patient is questioned about their fatigue and dyspnea levels using the Borg scale, and breaks are given when necessary. The aerobic exercise program is performed as a 12-week, 3-day-a-week self-walking exercise. The walking program is performed in the form of walking on flat ground at 60% workload, based on the data obtained from the 6-minute walking test result (land-based walking).
  Arms: Pulmonary Rehabilitation Group (PGr)
Genetic: No intervention — Peripheral blood samples will be taken once from the participants in the control group and no other intervention will be performed.
  Arms: Control Group (KGr)

SUMMARY:
The goal of this observational study is to examine the effects of traditional respiratory rehabilitation and respiratory muscle strengthening training added to this program at the genetic level in asthma. The main questions it aims to answer are:

* Does respiratory muscle strengthening exercise added to respiratory rehabilitation in asthmatic patients have additional benefits on rehabilitation outcome measures such as exercise capacity, shortness of breath, and muscle strength?
* Does the gain obtained with respiratory muscle strengthening in asthmatic patients increase the quality of life of patients and have a positive effect on their psychological state?
* Does respiratory rehabilitation applied to asthmatic patients have an effect on genetic changes?
* Does respiratory muscle strengthening training applied in addition to respiratory rehabilitation in asthmatic patients have an effect on genetic changes?
* Participants will be included in two different respiratory rehabilitation programs with and without respiratory muscle training, and pre- and post-treatment rehabilitation criteria and genetic changes will be compared.

DETAILED DESCRIPTION:
Asthma is the most common chronic respiratory disease worldwide, characterized by inflammation in the respiratory tract accompanied by bronchoconstriction, edema, and increased mucosa. Oxidative stress causes smooth muscle contraction, proliferation, and hypersensitivity of the airways, while hypoxia and systemic inflammation weaken the respiratory muscles. Lung hyperinflation in asthmatic patients causes an increase in the work of breathing. The increased workload on the respiratory muscles increases the respiratory frequency and causes dyspnea.

Pharmacological agents, allergen avoidance, lifestyle modification, anti-IgE antibodies and selectively alternative/complementary drugs or non-pharmacological methods (including breathing exercises, pulmonary rehabilitation, yoga and inspiratory muscle training) are applied in the treatment of asthma. Exercise training; it has been reported to improve asthma symptoms, quality of life, exercise capacity, bronchial hyperresponsiveness, exercise-induced bronchoconstriction and cardiopulmonary fitness and reduce airway inflammation and nighttime symptoms in asthmatic patients. In addition, asthma control can be increased with appropriate timing and intensity of exercise-based PR. The physiological effect of inspiratory muscle training is to weaken the metaboreflex mechanism, possibly reducing the activity of chemosensitive afferents and sympathetic nerve stimulation. Inspiratory muscle training stimulates structural and biochemical adaptations within the inspiratory muscles. It is stated in the literature that physiotherapy approaches such as breathing exercises and respiratory muscle training provide clinical benefits by increasing inspiratory muscle strength and reducing symptoms and the need for bronchodilators.

In recent years, the role of lncRNAs has also been emphasized in studies conducted on asthma patients. LncRNAs are long non-coding RNAs and there are studies indicating that they play an important role in the regulation of asthma. However, there is no study in the literature examining the effect of exercise training on lncRNA MALAT1 in asthmatic patients. Asthma is the most common chronic respiratory disease worldwide, characterized by inflammation in the respiratory tract accompanied by bronchoconstriction, edema, and increased mucosa. Oxidative stress causes smooth muscle contraction, proliferation, and hypersensitivity of the airways, while hypoxia and systemic inflammation weaken the respiratory muscles. Lung hyperinflation in asthmatic patients causes an increase in the work of breathing. The increased workload on the respiratory muscles increases the respiratory frequency and causes dyspnea.

Pharmacological agents, allergen avoidance, lifestyle modification, anti-IgE antibodies and selectively alternative/complementary drugs or non-pharmacological methods (including breathing exercises, pulmonary rehabilitation, yoga and inspiratory muscle training) are applied in the treatment of asthma. Exercise training; it has been reported to improve asthma symptoms, quality of life, exercise capacity, bronchial hyperresponsiveness, exercise-induced bronchoconstriction and cardiopulmonary fitness and reduce airway inflammation and nighttime symptoms in asthmatic patients. In addition, asthma control can be increased with appropriate timing and intensity of exercise-based PR. The physiological effect of inspiratory muscle training is to weaken the metaboreflex mechanism, possibly reducing the activity of chemosensitive afferents and sympathetic nerve stimulation. Inspiratory muscle training stimulates structural and biochemical adaptations within the inspiratory muscles. It is stated in the literature that physiotherapy approaches such as breathing exercises and respiratory muscle training provide clinical benefits by increasing inspiratory muscle strength and reducing symptoms and the need for bronchodilators.

In recent years, the role of lncRNAs has also been emphasized in studies conducted on asthma patients. LncRNAs are long non-coding RNAs and there are studies indicating that they play an important role in the regulation of asthma. However, there is no study in the literature examining the effect of exercise training on lncRNA MALAT1 in asthmatic patients. The research is a preliminary study for further studies in this field.Asthma is the most common chronic respiratory disease worldwide, characterized by inflammation in the respiratory tract accompanied by bronchoconstriction, edema, and increased mucosa. Oxidative stress causes smooth muscle contraction, proliferation, and hypersensitivity of the airways, while hypoxia and systemic inflammation weaken the respiratory muscles. Lung hyperinflation in asthmatic patients causes an increase in the work of breathing. The increased workload on the respiratory muscles increases the respiratory frequency and causes dyspnea.

Pharmacological agents, allergen avoidance, lifestyle modification, anti-IgE antibodies and selectively alternative/complementary drugs or non-pharmacological methods (including breathing exercises, pulmonary rehabilitation, yoga and inspiratory muscle training) are applied in the treatment of asthma. Exercise training; it has been reported to improve asthma symptoms, quality of life, exercise capacity, bronchial hyperresponsiveness, exercise-induced bronchoconstriction and cardiopulmonary fitness and reduce airway inflammation and nighttime symptoms in asthmatic patients. In addition, asthma control can be increased with appropriate timing and intensity of exercise-based PR. The physiological effect of inspiratory muscle training is to weaken the metaboreflex mechanism, possibly reducing the activity of chemosensitive afferents and sympathetic nerve stimulation. Inspiratory muscle training stimulates structural and biochemical adaptations within the inspiratory muscles. It is stated in the literature that physiotherapy approaches such as breathing exercises and respiratory muscle training provide clinical benefits by increasing inspiratory muscle strength and reducing symptoms and the need for bronchodilators.

In recent years, the role of lncRNAs has also been emphasized in studies conducted on asthma patients. LncRNAs are long non-coding RNAs and there are studies indicating that they play an important role in the regulation of asthma. However, there is no study in the literature examining the effect of exercise training on lncRNA MALAT1 in asthmatic patients. The research is a preliminary study for further studies in this field.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 75,
* Being diagnosed with severe persistent asthma by a chest physician in accordance with the Global Initiative for Asthma (GINA) guideline criteria,
* Patients with type 2 inflammation markers. According to the accepted standard; Peripheral eosinophils ≥150/µL and/or induced sputum eosinophils ≥2% - Airway hyperresponsiveness (PC20 methacholine < 8 mg/mL) and/or bronchodilator response (>12% or 200 mL improvement in % predicted FEV1 following 400 mg salbutamol inhalation)

Exclusion Criteria:

* Having had a recent (within the last month) respiratory tract infection,
* Having a smoking history of over 10 packs/years or having a smoking history within 6 months of quitting smoking,
* Having received oral corticosteroid treatment within the last 4 weeks,
* Having a Body Mass Index >30,
* Eosinophilic Granulomatosis with Polyangiitis (EGPA) and Allergic Bronchopulmonary Aspergillosis (ABPA),
* Vasculitis,
* History of malignancy,
* Pregnancy,
* Presence of a musculoskeletal, neurological or cardiac disease that would prevent exercise.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
lncRNA MALAT1 expression levels | Baseline and 12 weeks
  Real-time PCR will be performed twice for each sample for each gene, and after all the steps, ΔCT, ΔΔCT, 2^(ΔΔCT) fold change in expression between the experiment and control.
Respiratory Muscle Strength Measurement | Baseline and 12 weeks
  The patient is seated in a straight-backed chair. The patient is asked to grasp the silicone mouthpiece with his/her mouth and inhale and exhale as quickly and deeply as possible. The measurements are repeated until 3 measurement values are obtained with a maximum of 10% deviation between the measured peak value. The maximum value is taken among the measured values.
Forced Expiratory Volume in 1 s (FEV1 ) | Baseline and 12 weeks
  FEV1 will perform by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines.
Exercise capacity | Baseline and 12 weeks
  A 6-minute walk test is performed for exercise capacity. After resting in a chair for a sufficient period (>30 minutes), patients walk as fast as possible, without running, for 6 minutes on a straight 30-meter corridor. Before and after the test, the patient's fatigue and dyspnea are questioned using the Modified Borg Scale. Oxygen saturation and heart rate are monitored and recorded using a finger pulse oximeter before, during, and after the test.
Forced Vital Capacity (FVC) | Baseline and 12 weeks
  FVC will perform by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines.
FEV1/FEVC | Baseline and 12 weeks
  FEV1/FEVC will perform by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines.

SECONDARY OUTCOMES:
Asthma Control Test (ACT-ACQ) | Baseline and 12 weeks
  ACQ is a scale that evaluates the patient's perspective on their current asthma control level, which can be used to evaluate the general status of their asthma control. The test consists of five questions, the highest score is 25 and the lowest score is zero. A score of 25 indicates full control, while a score between 24-20 indicates partial control. A score below 19 on the scale indicates that asthma is uncontrolled.
Asthma Quality of Life Scale (AQLQ) | Baseline and 12 weeks
  It is a 32-question asthma-specific quality of life scale. It evaluates the responses with a 7-point scale (1: Severe effect, 7: No effect). It consists of 12 different questions about asthma symptoms, 11 about activity limitation, 5 about emotional function and 4 about environmental factors. Total score average and average scores for sub-dimensions are calculated.
Modified Medical Research Council (mMRC) Dyspnea Scale | Baseline and 12 weeks
  mMRC is a 0-4 point category scale where patients select the value that best describes their level of dyspnea. Increases in mMRC levels, especially values of 2 and above, are considered to indicate an increased risk of mortality.
International Physical Activity Questionnaire-Short form (IPAQ-SF) | Baseline and 12 weeks
  It is an internationally valid questionnaire for the assessment of physical activity. The short form of the questionnaire consists of seven questions and provides information about the time spent in sitting, walking, moderate and intense activities. A score is obtained as "MET-minutes/week" by multiplying minutes, days and MET values. The numerical values obtained are classified as inactive, minimally active or very active.
Digital muscle strength measurement | Baseline and 12 weeks
  Muscle strength is assessed using an electronic hand dynamometer. The patient is asked to maintain muscle strength against the dynamometer for at least 5 seconds in each attempt, with the force measurement repeated 3 times. The best value from the 3 test results is recorded.
Hospital Anxiety and Depression Scale (HADS) | Baseline and 12 weeks
  It is a scale that questions whether patients have clinical symptoms of anxiety and depression. HADS-A is the anxiety subscale and consists of 7 questions, while HADS-D is the depression subscale and consists of 7 questions. Scoring is between 0-21 for both tests. An increase in the score on the scale means that the severity of anxiety and depression increases. The cut-off points were 10 for the anxiety subscale and 7 for the depression subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Esra PEHLİVAN, Assoc. Prof., Study Chair — Saglik Bilimleri Universitesi; Erdoğan ÇETİNKAYA, Prof. Dr., Study Director — Yedikule Chest Diseases And Thoracic Surgery Training And Research Hospital; Fulya Senem KARAAHMETOGLU, PhD (c), Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No